CLINICAL TRIAL: NCT00644371
Title: Allogeneic Transplantation of Haematopoietic Stem Cells Following Non-myeloablative Conditioning With Melphalan, Fludarabine, Thiotepa, Rituximab and Ibritumomab Tiuxetan (Zevalin) in Patients With Aggressive Non-Hodgkin's B-cell Lymphoma
Brief Title: Allogenic Stem Cell Transplantation (SCT) With Non-myeloablative Conditioning in Patients With Relapse Non-Hodgkin's Lymphoma (NHL)
Acronym: Z-RIC-Allo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO-Z-RIC-Allo; EuDRACT nº:2007-003302-10
Record Dates: First submitted 2008-03-18; First posted 2008-03-26 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Allogeneic; Lymphoma; GELTAMO; Z-RIC
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Ibritumomab Tiuxetan (Zevalin)

INTERVENTIONS:
Drug: Ibritumomab Tiuxetan (Zevalin) — Conditioning Regimen
  1. Rituximab, 250 mg/m2 on days -21 and -14.
  2. Ibritumomab tiuxetan (Zevalin): 0.4 mCi/kg (14.8 MBq/kg). Maximum: 32 mCi on day -14.
  Chemotherapy:
  * Fludarabine 30 mg/m2/day on days -7, -6, -5, -4 and -3 as a 30-min infusion.
  * Melphalan 70 mg/m2/day on days -3 and -2 as a 15-min infusion.
  Chemotherapy for relapsing patients after autologous transplantation including melphalan over the last 6 months:
  * Thiotepa 5 mg/kg over 4 hours every 12 hours on day -8.
  * Fludarabine 30 mg/m2/day on days -7, -6, -5, -4 and -3 as a 30-min infusion.
  * Melphalan 70 mg/m2/day on day -2 as a 15-min infusion.
  Other Names: Rituximab (Mabthera)

SUMMARY:
To evaluate the use of ibritumomab tiuxetan (Zevalin) as part of the non myeloablative conditioning with melphalan, fludarabine and thiotepa in patients submitted to allogeneic transplantation of haematopoietic stem cells from family donor's peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histologically confirmed B-cell lymphoma of the following subtypes:

   * LBCDL
   * Grade 3b follicular lymphoma
   * Mantle-cell lymphoma
   * Transformed B-cell lymphoma
   * Burkitt lymphoma in patients not eligible for a conventional allogeneic transplant
3. High-risk B-cell CD20+ lymphoma defined by

   * Having attained less than PR after two chemotherapy lines
   * Post-transplantation relapse
   * Presence of disease detected through a metabolic approach (PET/CT or else CT+PET) either before or after autologous transplantation
   * Inability to collect enough stem cells for autologous transplantation
4. Stable disease at the time of transplantation
5. Age between 18 and 65
6. Performance status (ECOG) ≤ 2
7. Normal and suitable pulmonary function (DLCO ≥ 30%)
8. Left ventricular ejection fraction (LVEF) determined by ventriculography or echocardiogram ≥ 40%
9. Normal hepatic and renal function, with creatinine ≤ 2 mg/dl and Bi ≤ 1.5 mg/dl, and alkaline phosphatase ≤ 2.5 x UNL ; AST, ALT ≤ 2.5 x UNL (≤ 5 x UNL if hepatic infiltration)

Exclusion Criteria:

1. Prior treatment with radiopharmaceutical agents
2. HIV-associated lymphoma
3. Presence of human anti-mouse antibodies (HAMA) or anti-chimeric antibodies (HACA)
4. Patient's inability to follow the protocol
5. Hypersensitivity to 90Y-itritumomab tiuxetan
6. Presence of severe pathologies that preclude chemotherapeutic treatment
7. Pregnant women or pregnancy risk due to inappropriate contraceptive measures
8. Breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02-21 (Actual); Study Completion 2013-02-04 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 12 months

SECONDARY OUTCOMES:
safety (toxicity, transplantation- and graft-related mortality) | 36 months
response to treatment according to the Cheson's criteria (Cheson B, et al. JCO 25, 570, 2007). | 36 months
overall survival | 36 months
relapse rate | 36 months
acute and chronic Graft-versus-Host Disease | 36 months
haematological and immunological reconstitution, and chimerism. | Post transplantation. Once weekly until day +100 and every 2 weeks from day +100.
the impact of Complete Clinical Response, determined by flow cytometry and PET, on progression-free survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Caballero, MD, Principal Investigator — Hospital Clínico Universitario de Salamanca
Locations (14):
- Spain (14):
  - H. Santa Creu i Sant Pau., Barcelona, Barcelona.
  - H. U. Marqués de Valdecilla., Santander, Cantabria
  - H.U. 12 de Octubre, Madrid, Madrid
  - H.U. Gregorio Marañón, Madrid, Madrid
  - H.U. La Princesa, Madrid, Madrid
  - H.U. Ramón y Cajal., Madrid, Madrid
  - H. Morales Meseguer., Murcia, Murcia
  - H. Virgen de la Arrixaca, Murcia, Murcia
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - H. Central de Asturias, Oviedo, Oviedo
  - H. Clinico de Salamanca, Salamanca, Salamanca
  - H. Clínico Valencia, Valencia, Valencia
  - H. La Fe, Valencia, Valencia
  - H.U. Miguel Servet, Zaragoza, Zaragoza.

REFERENCES:
- [Derived] Cabrero M, Martin A, Briones J, Gayoso J, Jarque I, Lopez J, Grande C, Heras I, Arranz R, Bernal T, Perez-Lopez E, Lopez-Godino O, Conde E, Caballero D. Phase II Study of Yttrium-90-Ibritumomab Tiuxetan as Part of Reduced-Intensity Conditioning (with Melphalan, Fludarabine +/- Thiotepa) for Allogeneic Transplantation in Relapsed or Refractory Aggressive B Cell Lymphoma: A GELTAMO Trial. Biol Blood Marrow Transplant. 2017 Jan;23(1):53-59. doi: 10.1016/j.bbmt.2016.10.003. Epub 2016 Oct 19. PMID 27771496